CLINICAL TRIAL: NCT02238847
Title: Randomized Controlled Trial Comparing Covered and Uncovered Biliary Self Expanding Metal Stents (SEMS) for Pre-operative Drainage During Neoadjuvant Therapy in Patients With Pancreatic Cancer
Brief Title: Pre-operative Biliary SEMS RCT During Neoadjuvant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90905950; E7034 (Other: Boston Scientific)
Record Dates: First submitted 2014-05-02; First posted 2014-09-12 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; Pancreatic Cancer; Preoperative Biliary Drainage; Neoadjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WallFlex Biliary RX Fully Covered Stent System (Active Comparator): Patients in this group will receive a fully covered study SEMS (self-expanding metal stent)
  Reintervention can occur with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System
  Interventions: Device: WallFlex™ Biliary RX Fully Covered/Uncovered Stent System
- WallFlex Biliary RX Uncovered Stent System (Active Comparator): Patients in this group will receive an uncovered study SEMS (self-expanding metal stent).
  Reintervention can occur with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System
  Interventions: Device: WallFlex™ Biliary RX Fully Covered/Uncovered Stent System

INTERVENTIONS:
Device: WallFlex™ Biliary RX Fully Covered/Uncovered Stent System — Reintervention can occur in Arm 1 or Arm 2 with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of Fully Covered biliary SEMS to Uncovered biliary SEMS in biliary drainage for the pre-operative management of biliary obstructive symptoms caused by pancreatic cancer in patients undergoing neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patient indicated for biliary metal stent placement for the treatment of jaundice and/or cholestasis
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study
* Suspicion of pancreatic adenocarcinoma
* Likely indicated for neoadjuvant treatment
* Distal biliary obstruction consistent with pancreatic cancer
* Location of distal biliary obstruction such that it would allow the proximal end of a stent to be positioned at least 2 cm from the hilum
* Endoscopic and surgical treatment to be provided at the same institution

Exclusion Criteria:

* Benign biliary strictures
* Malignancy secondary to Intraductal Papillary Mucinous Neoplasm
* Surgically altered anatomy where ERCP is not possible
* Previous biliary drainage using a SEMS or multiple plastic stents
* Contraindications for endoscopic techniques
* Patients who are currently enrolled in another investigational trial that would directly interfere with the current study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yousuke Nakai, MD, PhD, Principal Investigator — Tokyo University; Dong-Wan Seo, MD, Principal Investigator — Asan Medical Center
Locations (9):
- United States (4):
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- CUB Hopital Erasme, Brussels, Belgium
- Centre Hospitalier de l'Université de Montréal-Saint-Luc Hospital, Montreal, Quebec, Canada
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy
- Tokyo University Hospital, Tokyo, Japan
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Seo DW, Sherman S, Dua KS, Slivka A, Roy A, Costamagna G, Deviere J, Peetermans J, Rousseau M, Nakai Y, Isayama H, Kozarek R; Biliary SEMS During Neoadjuvant Therapy Study Group. Covered and uncovered biliary metal stents provide similar relief of biliary obstruction during neoadjuvant therapy in pancreatic cancer: a randomized trial. Gastrointest Endosc. 2019 Oct;90(4):602-612.e4. doi: 10.1016/j.gie.2019.06.032. Epub 2019 Jul 2. PMID 31276674

RESULTS

PARTICIPANT FLOW:
Groups:
- WallFlex Biliary RX Fully Covered Stent System: Patients in this group will receive a fully covered study SEMS (self-expanding metal stent)
  Reintervention can occur with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System
  WallFlex™ Biliary RX Fully Covered/Uncovered Stent System: Reintervention can occur in Arm 1 or Arm 2 with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System
- WallFlex Biliary RX Uncovered Stent System: Patients in this group will receive an uncovered study SEMS (self-expanding metal stent).
  Reintervention can occur with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System
  WallFlex™ Biliary RX Fully Covered/Uncovered Stent System: Reintervention can occur in Arm 1 or Arm 2 with either a WallFlex™ Biliary RX Fully Covered or Uncovered Stent System
Period: Overall Study
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Started | 59 | 60
Completed | 37 | 36
Not Completed | 22 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [58.0 to 71.0] | 65.0 [58.5 to 73.0] | 65 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 33 | 33 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Median (Inter-Quartile Range); unit: kg] | 77.7 [62.3 to 87] | 78.4 [65.1 to 90.4] | 78 [64.6 to 89.9]
Gallbladder in Situ [Count of Participants; unit: Participants] — A count of participants with no prior history of cholecystectomy (gallbladder still in place).
  Participants | 43 | 42 | 85
Karnofsky Score (overall health status) [Median (Inter-Quartile Range); unit: units on a scale] — 100 Normal no complaints nor evidence of disease;90 Normal activity, minor signs/symptoms of disease;80 Normal activity w/effort, some sign/symptom of disease;70 Cares for self, unable to carry on normal activity/do active work;60 Requires occasional assistance, able to care for most personal needs;50 Requires considerable assistance & frequent medical care;40 Disabled, requires special care/assistance;30 Severely disabled, hospitalization indicated, death not imminent;20 Very sick, hospitalization & active support treatment necessary;10 Moribund, fatal processes progress rapidly;0 Dead
  units on a scale | 90.0 [80.0 to 100.0] | 80.0 [80.0 to 90.0] | 90 [80 to 90]
Tumor Size [Mean (Standard Deviation); unit: cm] | 3.1 (1.4) | 2.9 (50.9) | 3.0 (1.2)
Tumor Stage [Count of Participants; unit: Participants] — Tumor, Node, Metastasis Cancer Staging System:
  Primary Tumor (T)1-4: Tumor size and extent; higher number indicates larger tumor and/or spread to nearby tissues Regional Lymph Node (N)0-3: N0 no regional lymph node involvement; 1-3 indicates number of regional lymph nodes involved and extent of involvement (higher number is more lymph node involvement) Distant Metastasis (M)0: No distant metastases
  Participants
    IA - T1 N0 M0 | 7 | 3 | 10
    IB - T2 N0 M0 | 5 | 6 | 11
    IIA - T3 N0 M0 | 19 | 24 | 43
    IIB - T1 N1 M0; T2 N1 M0; T3 N1 M0 | 15 | 15 | 30
    III - T4 Any N M0 | 5 | 5 | 10
    Unknown | 8 | 7 | 15
Number of participants who underwent curative intent surgery [Count of Participants; unit: Participants] | 24 | 27 | 51
Number of participants not undergoing curative intent surgery&followed to 1year post-stent placement [Count of Participants; unit: Participants] | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Sustained Biliary Drainage, Defined as Absence of Reinterventions for the Management of Biliary Obstructive Symptoms
Description: Sustained biliary drainage, defined as absence of reinterventions for the management of biliary obstructive symptoms, assessed from self-expanding metal stent (SEMS) placement until curative intent surgery (CIS) when applicable, or to one year after SEMS placement otherwise.
Time Frame: From SEMS placement until CIS (for patients undergoing CIS; median 110 days to CIS) or from SEMS placement to one year after SEMS placement (for patients not undergoing CIS)
Population: Participant was eligible for primary endpoint analysis if participant did not undergo biliary reintervention from time of SEMS placement to CIS, or from time of SEMS placement to one year after SEMS placement (for participants not undergoing CIS).
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 54 | 59
Participants | 39 | 43
Statistical Analysis 1: Comparison: WallFlex Biliary RX Fully Covered Stent System vs WallFlex Biliary RX Uncovered Stent System; Test type: Non-Inferiority — The prespecified non-inferiority margin was set at 20%. This was chosen to support a practical study size while still able to identify major differences if this were the case; p < 0.01, Exact Non-inferiority — Reported p-value of <0.01 is calculated p-value. (p<0.05 was considered significant)

2. Secondary Outcome: Procedure-related or Stent-related Serious Adverse Events
Description: Serious adverse events related to the stent placement procedure or to the stent
Time Frame: From stent placement procedure up to one year after stent placement procedure
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 59 | 60
Participants | 14 | 12
Statistical Analysis 1: Comparison: WallFlex Biliary RX Fully Covered Stent System vs WallFlex Biliary RX Uncovered Stent System; Test type: Superiority; p = 0.66, Fisher Exact

3. Secondary Outcome: Technical Success
Description: Technical success defined as the ability to deploy the stent in a satisfactory position across the stricture; proximal end of the stent is no more than 1-2cm beyond the proximal end of the stricture.
Time Frame: During the Stent Placement Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 59 | 60
Participants | 58 | 60

4. Secondary Outcome: Ability to Complete Neoadjuvant Therapy as Intended Without Stent-related Interruptions of Neoadjuvant Therapy and Without Biliary Reintervention
Description: The ability to complete neoadjuvant therapy as intended without stent-related interruptions of neoadjuvant therapy and without biliary reintervention
Time Frame: From initial stent placement procedure to curative intent surgery (CIS) (median 110 days to CIS), or from initial stent placement procedure to one year after initial stent placement for participants not undergoing CIS
Population: Of 59 participants in the Fully Covered arm, neoadjuvant therapy information was only provided for 55 participants. Of 60 participants in the Uncovered arm, neoadjuvant therapy information was only provided for 52 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 55 | 52
Participants | 53 | 51

5. Secondary Outcome: Number of Participants With Stent Migration
Description: The number of participants with stent migration
Time Frame: At the time of curative intent surgery (CIS) (median 110 days to CIS) or transition to palliation for participants not underoing CIS
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 59 | 60
Participants | 5 | 0

6. Secondary Outcome: Subjective Impression of the Surgeon That the Presence of a Self-expanding Metal Stent May Have Impacted the Surgical Procedure
Description: The subjective impression of the surgeon that the presence of a self-expanding metal stent (SEMS) may have impacted the surgical procedure.
Time Frame: At the time of curative intent surgery (CIS) (median 110 days to CIS)
Population: Of 59 Participants in Fully Covered Arm, 24 underwent Curative Intent Surgery. Of 60 Participants in Uncovered Arm, 27 underwent Curative Intent Surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 24 | 27
Participants | 3 | 4

7. Secondary Outcome: For Participants Not Undergoing Curative Intent Surgery, Sustained Biliary Drainage to One Year After Stent Placement
Description: For participants not undergoing curative intent surgery, sustained biliary drainage from stent placement to one year after stent placement.
Time Frame: From stent placement to one year after stent placement for participants not undergoing curative intent surgery
Population: 30 participants in the Fully Covered arm did not undergo curative intent surgery and were followed for one year. 32 participants in the Uncovered arm did not undergo curative intent surgery and were followed for one year.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 30 | 32
Participants | 19 | 21

8. Post Hoc Outcome: Number of Participants With Tumor Ingrowth
Description: The number of participants with tumor ingrowth at any point during stent indwell.
Time Frame: Measured at any point during stent indwell - until curative intent surgery (CIS) (median 110 days to CIS) or one year post stent placement (for participants not underoing CIS)
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 59 | 60
Participants | 0 | 10

9. Post Hoc Outcome: Number of Participants With Acute Cholecystitis
Description: The number of participants with acute cholecystitis
Time Frame: From stent placement up to curative intent surgery (CIS) (median 110 days to CIS), or from stent placement up to one year post stent placement for participants not undergoing CIS
Population: 43/59 participants in Fully Covered Arm and 42/60 participants in Uncovered Arm had gallbladder in situ. Therefore, Acute Cholecystitis only analyzed in 43 participants in Fully Covered Arm and 42 participants in Uncovered Arm.
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 43 | 42
Participants | 4 | 2

10. Post Hoc Outcome: Mortality at One Year After Randomization
Description: The mortality at one year after randomization.
Time Frame: From randomization to one year after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
Number analyzed (Participants) | 59 | 60
Participants | 21 | 25

ADVERSE EVENTS:
Time Frame: Adverse event data collected from the time the participant signed the informed consent and was randomized to the study, to the time the participant exited the study (median of 344 days of follow-up).
Description: Reported on all treatment related Serious Adverse Events
Arm/Group | WallFlex Biliary RX Fully Covered Stent System | WallFlex Biliary RX Uncovered Stent System
All-Cause Mortality (participants affected / at risk) | 21/59 | 25/60
Serious Adverse Events (participants affected / at risk) | 14/59 | 12/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WallFlex Biliary RX Fully Covered Stent System (N=59) | WallFlex Biliary RX Uncovered Stent System (N=60)
Acute Cholecystitis (Hepatobiliary disorders) | 4 | 2
Acute Pancreatitis (Gastrointestinal disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 9 | 8
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
CBD Obstruction or Abnormal LFTs (Hepatobiliary disorders) | 2 | 1
Liver Abscess (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02238847/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT02238847/SAP_001.pdf